CLINICAL TRIAL: NCT05641051
Title: Effects of Metoclopramide Administration on Gastric Emptying in Mechanically Ventilated Critically Ill Patients : A Prospective Randomized Controlled Trial
Brief Title: Metoclopramide on Gastric Emptying in Mechanically Ventilated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Mohammed Elbaradei, Resident of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 35298/2/22
Record Dates: First submitted 2022-11-27; First posted 2022-12-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Gastric Emptying; Mechanically Ventilation; Randomized Controlled Trial; Metoclopramide
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The drugs will be prepared by a dedicated anesthesiologist who is aware of the allocated group and will have no subsequent role in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoclopramide group (Experimental): Patients will receive 10 mg intravenous metoclopramide / 6 hours.
  Interventions: Drug: Metoclopramide
- Control group (Placebo Comparator): Patients will receive the same volume of intravenous placebo / 6 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — Cases will receive 10 mg intravenous metoclopramide every 6 hours.
  Arms: Metoclopramide group
Drug: Placebo — Cases will receive the same volume of IV placebo / 6 hours.
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the prokinetic effect of metoclopramide on gastric emptying in critically ill mechanically ventilated patients .

DETAILED DESCRIPTION:
More than 50% of patients in ICU have gastric dysmotility, which leads to slow gastric emptying(GE) and high gastric residual volume (GRV) and is associated with increased mortality in these patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age 20 - 60 years.
2. Either gender.
3. Mechanically ventilated head trauma patients.
4. Patients receiving enteral feeding via nasogastric tube.

Exclusion Criteria:

1. Patients with contraindications to enteral feeding.
2. Patients with extrapyramidal manifestations.
3. Patients with known allergy to metoclopramide.
4. Patients with seizures.
5. Patients with renal or hepatic diseases.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Assessment of the risk of aspiration | 8 hours interval during first 5 days of enteral feeding
  Aspiration risk will be categorized using the system proposed by Ven de Putte and Perlas. As:
  * patients with empty antrum and gastric residual volume < 1.5 mL/kg: low risk.
  * patients with solid contents or gastric residual volume > 1.5 mL/kg: high risk.

SECONDARY OUTCOMES:
Incidence of ventilator associated pneumonia | 8 hours interval during first 5 days of enteral feeding
  Pneumonia will be defined according to the ATS/IDSA clinical criteria and will be diagnosed if a new or progressive radiographic infiltrate is present and at least two of the three following clinical features are also present: (1) fever higher than 38°C, (2) leukocytosis or leucopenia and (3) purulent secretions. No microbiological confirmation is required for diagnosis of pneumonia.
  Infectious Diseases. Society of America (IDSA) and the American Thoracic. Society (ATS)
Time of weaning from mechanical ventilation | From the start of enteral feeding till intensive care discharge through study completion, an average of 6months
  Time of weaning from mechanical ventilation From the start of enteral feeding
Hospital stay | From the start of enteral feeding till intensive care discharge through study completion, an average of 6months
  Hospital stay including intensive care and ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP